CLINICAL TRIAL: NCT06895096
Title: Comparison of Retention of Self-etch Sealants and Flowable Composite in Permanent Molars
Status: Completed | Type: Observational
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Shoaib Rahim, Associate Professor, Foundation University Islamabad
Other Study IDs: FUCDCLINIC-2407
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Pits and Fissures Sealant
Keywords: flowable composite; self-etch sealant; sealant retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 06 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Retention of self-Etch sealants vs flowable composite in contralateral molars: Comparison of retention of self-etch sealants and flowable composite in inter-arch contralateral molars
  Interventions: Device: Pit Fissure Sealant

INTERVENTIONS:
Device: Pit Fissure Sealant — Flowable composite is being used for the purpose of sealing pits and fissures which require etching and bonding before application whereas self etch sealants are self adhesive and do not require etching and sealing.

SUMMARY:
Comparison of Retention of Self-etch sealants and Flowable Composite in permanent Molars.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 8 to 18 years.
2. Patients with completely erupted maxillary and mandibular molars with deep pits and fissures having a score of 0 or 1 according to ICDAS classification -

Exclusion Criteria:

1. Patients with a history of any medical conditions such as Sjogren's syndrome , renal failure or have immunocompromised state (juvenile diabetes).
2. Patients with history of prolonged medication such as steroids, chemotherapy or TB medication.
3. Teeth with carious lesion extending to dentino-enamel junction/dentin.
4. Patients with poor oral hygiene.
5. Patients with bruxism or parafunctional habits.
6. Permanent molars with developmental defects or restorations.
7. Teeth with poor prognosis and having periodontal diseases.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients reporting to Paedodontics and Operative dentistry department of FUCD&H will be selected according to inclusion criteria after history, clinical examination & radiographic evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
sealant retention | from enrollment to end of treatment at 6 months
  observation as to whether sealant is completely retained ,partially retained or completely lost

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation university college of Dentistry and Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh C, Kaur K, Kapoor K. Retention of pit and fissure sealant versus flowable composite: An in vivo one-year comparative evaluation. J Indian Soc Pedod Prev Dent. 2019 Oct-Dec;37(4):372-377. doi: 10.4103/JISPPD.JISPPD_122_19. PMID 31710012
- See also: Retention of pit and fissure sealant versus flowable composite: An in vivo one-year comparative evaluation — https://pubmed.ncbi.nlm.nih.gov/31710012/